CLINICAL TRIAL: NCT00958100
Title: Phase IIb Pilot Study for the Evaluation of the Safety and the Feasibility of Treatment Simplification to Tenofovir+Emtricitabine+Raltegravir or to Lamivudine+Abacavir+Raltegravir in Patients With Optimal Virological Control and Toxicity to the Current Combined Antiretroviral Regimen
Brief Title: Raltegravir Switch for Toxicity or Adverse Events
Acronym: RaSTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Simona Di Giambenedetto, Dr, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-014316-35
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: HIV/AIDS; Antiretroviral Therapy; HIV Infections
Keywords: raltegravir switch toxicity; treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tenofovir Emtricitabine Raltegravir (Experimental): Patients switching to raltegravir with tenofovir+emtricitabine as backbone
  Interventions: Drug: tenofovir emtricitabine raltegravir
- Lamivudine Abacavir Raltegravir (Experimental): Switch from current antiretroviral regimen to raltegravir with abacavir/lamivudine as backbone
  Interventions: Drug: Lamivudine Abacavir Raltegravir
- Abacavir free (Experimental): Patients switched to raltegravir whose backbone therapy should not be randomized in order to avoid the use of abacavir (HLA-B*5701 positive patients,Framingham score 20% or higher)
  Interventions: Drug: Abacavir free

INTERVENTIONS:
Drug: tenofovir emtricitabine raltegravir — switch from current antiretroviral regimen to raltegravir with tenofovir/emtricitabine as backbone
  Arms: Tenofovir Emtricitabine Raltegravir
Drug: Lamivudine Abacavir Raltegravir — Switch from current antiretroviral regimen to raltegravir with abacavir/lamivudine as backbone
  Arms: Lamivudine Abacavir Raltegravir
Drug: Abacavir free — Patients will receive raltegravir with tenofovir/emtricitabine; data will be added to those of Tenofovir Emtricitabine Raltegravir arm in a separate longitudinal analysis comparing data at baseline and at 48 weeks. In this separate analysis, data will not be compared to those obtained from the Lamivudine Abacavir Raltegravir arm. The number of patients in this arm is not pre-established.
  Arms: Abacavir free

SUMMARY:
This study aims to verify the persistent control of the virus replication at 48 weeks after the simplification to tenofovir + emtricitabine + raltegravir or to lamivudine+abacavir+raltegravir in patients with optimal virological suppression without any virological failure to previous combined antiretroviral therapies needing a therapeutic switch for toxicity related issues or adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with a combined antiretroviral therapy from at least 1 year
* Aged 18 years or older
* With one or more of the following conditions:

  * Grade 3 or 4 Dyslipidemia
  * Any Hyperglycemia
  * Lipodystrophy (patient's self report, confirmed by physician's physical examination)
  * Moderate/severe cardiovascular risk, defined as a calcium score higher than 40 or a Framingham score higher than 10 (estimated 10 years cardiovascular risk: 10%)
  * Diarrhea (at least 3 emissions of loose stool every day for at least 3 days every week)
* With at least two HIV-RNA levels <50 copies/mL on two consecutive determinations at least 3 months apart
* With CD4 cell count >200 cells/ μL for at least 6 months and absence of any opportunistic infection or AIDS-related disease during the last year before screening.
* Who gave informed consent to the participation to the study

Exclusion Criteria:

* Pregnancy or breast feeding, desire of pregnancy in the short term
* Previous virological failure (two consecutive HIV-RNA levels > 50 copies/mL or a single value >1000 copies/mL) to antiretroviral therapy and/or previous exposure to mono- or dual therapies with reverse transcriptase nucleoside analogues except for patients with subsequent genotypic resistance tests showing no resistance mutations to any of the study drugs.
* Previous exposure to inhibitors of HIV-1 integrase
* Previous major toxicity to any of the study drugs
* Spontaneous treatment interruptions in disagreement with the treating physician in the last year or loss to follow-up for at least 6 months, at least once in the last two years
* Current alcohol or drug abuse or any other condition which, in the judgment of the treating physician, may impair the patient's adherence to the new drug regimen and/or to the protocol's procedures
* Patients with grade 3 or 4 laboratory abnormalities at screening (except for lipid and glucose levels)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To verify the persistent control of the virus replication after the simplification to tenofovir+emtricitabine+raltegravir or to lamivudine+abacavir+raltegravir in patients with optimal virological suppression without any previous virological failure | 48 weeks

SECONDARY OUTCOMES:
Time to virological failure (two consecutive HIV-RNA levels > 50 copies/mL or a single value >1000 copies/mL) at survival analysis | 48 weeks
Proportion of patients with viral load lower than 50 copies/mL at 48 weeks at the intention to treat analysis | 48 weeks
Evolution of CD4 cell count during the 48 weeks of study | 48 weeks
Evolution of adherence and quality of life during the 48 weeks of study | 48 weeks
Evolution of raltegravir plasma concentrations during the 48 weeks of study | 48 weeks
Evolution of metabolic parameters during the 48 weeks of study | 48 weeks
Change of the results of neurocognitive tests at 48 weeks of study | 48 weeks
Change of bone density and of adipose tissue by DEXA analysis at 48 weeks of study | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico A. Gemelli, Rome, Italy